CLINICAL TRIAL: NCT02851862
Title: A Natural History of Late Onset Tay-Sachs Disease: MGH Site
Brief Title: A Natural History of Late Onset Tay-Sachs Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Florian Eichler, Director of the Center for Rare Neurological Diseases, Massachusetts General Hospital
Other Study IDs: 2015P002399
Record Dates: First submitted 2016-07-19; First posted 2016-08-02 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: GM2 Gangliosidosis
MeSH Terms: conditions — Gangliosidoses, GM2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood will be collected to establish lymphoblast cell lines. Cerebrospinal fluid will also be collected from some subjects.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Late Onset GM2 Gangliosidosis: 10-15 subjects with Late Onset GM2 Gangliosidosis

SUMMARY:
The purpose of this study is to learn more about the natural history of Late Onset GM2 Gangliosidosis (Tay-Sachs disease and Sandhoff Disease) to inform future clinical trials.

DETAILED DESCRIPTION:
For this study, subjects will come to Massachusetts General Hospital for two study visits, six months apart. At each visit, the following tests will be done:

A Neurological Exam, Several Ataxia Rating Scales, A Formal Speech assessment, Magnetic resonance imaging and spectroscopy, A blood draw, An optional lumbar puncture.

Outcome measures and biomarkers (MRI atrophy measures, chemical shift imaging (CSI), MRS and CSF metabolites) will be compared to the clinical disease course in Late Onset GM2 Gangliosidosis. The natural history by retrospective surveys (previously acquired) will shed light on how changes in outcome measures compare to the larger context of changing symptoms (that occurs on the scale of years and decades). This combined approach will elucidate optimal outcome measures and determine eligibility criteria for a future clinical trial in Late Onset GM2 Gangliosidosis.

The international web-based platform for clinical research networks, NeuroBANK™, in which clinicians and researchers collect and share their patients' clinical and research data, will be used. This system has been implemented by and deployed at the Neurological Clinical Research Institute at Massachusetts General Hospital. This platform allows clinicians to enter patient data, either a) manually via a Web-based interface, or b) by exporting the data from the electronic health record (EHR) and clinical data repositories.

VIDEO OCULOGRAPHY:

Eye movement analysis will be performed in some patients using a formal video oculography setup jointly with a portable setup. The findings will be assessed to see if respective assessments concur.

GLOBAL UNIQUE IDENTIFIERS (GUID):

A patient Global Unique Identifier (GUID) will be used as the identifier for individuals participating in the study in NeuroBANK™. The GUID is an 11-character string that is generated using encryption technology and algorithms licensed by the NCRI from the National Institutes of Health (NIH).

The GUID is generated on a secure website that utilizes 128-bit Secure Socket Layer (SSL). Of note, this website is not linked to NeuroBANK™. The GUID is generated using an irreversible encryption algorithm - it accepts twelve identifying data elements, (e.g. last name at birth, first name at birth, gender at birth, day, month and year of birth, city and country of birth, etc.), and produces a unique random-generated character string, or GUID. No identifying information is stored in the system; it is simply used to generate the GUID. If the same information is entered again, the same GUID will be returned.

The GUID is entered into NeuroBANK™ when the patient is being created in the system. As the same patient may participate in multiple studies, NeuroBANK™ will also allow capturing a study-specific ID for the patient. For more information about NeuroBANK™ or the GUID, please go to: www.neurobank.org.

Data Management:

The NCRI Data Management Team is trained and knowledgeable regarding confidentiality and integrity of data. They will be responsible for all aspects of data procedures. Alex Sherman is the ALD Connect network strategist and member of the NEALS ALS consortium. He is the director of Strategic Development and Systems of NCRI, serves on the Executive Committee of the ALS Research Group, and is one of the leaders of the NEALS ALS Consortium.

Data Quality Checks, Logic Checks and Queries:

The Data Manager (DM) at the Neurological Clinical Research Institute (NCRI) at the Massachusetts General Hospital will conduct monthly Data Quality Checks, Logic Checks, and internal data quality audits. Data field queries will be resolved in an established workflow according to the Standard Operating Procedures (SOPs). The queries may be created either at the point of entry during the data entry process, manually by the NCRI DM, or as the result of executing monthly Logic Checks.

Study-Specific Database Backup and Maintenance:

The NCRI personnel will be responsible for the database backups that will be conducted daily. Simultaneously, a separate copy of the backup in the encrypted compressed format will be maintained and saved by the System Analysts. The backups will be saved on a separate computer partition in a password-protected compressed format and also will be burnt into DVD medium and stored in a secure location.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have a confirmed diagnosis of Late Onset GM2 Gangliosidosis as defined by (a) absent to near-absent beta-hexosaminidase enzymatic activity in the serum or white blood cells or (b) mutation analysis of the HEXA and HEXB genes to distinguish pseudo deficiency alleles from disease-causing alleles
* The subject must be older than 7 years of age

Exclusion Criteria:

* If a patient is very severely affected by the disease, the PI will assess whether it is in the best interest of the patient to exclude them from the study for their own comfort and well being. In cases where the PI deems it appropriate, severely affected patients will be excluded. Patients under the age of 7 years will be excluded from this study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects diagnosed with Late Onset GM2 Gangliosidosis
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Ataxia Rating Scale over six months | baseline and 6 month visits
  Ataxia rating scale incorporating gait, dysarthria, and coordination

SECONDARY OUTCOMES:
Change over six months in metabolite levels seen on magnetic resonance spectroscopy | baseline and 6 months
  Metabolite levels
Change over six months in lipid levels found in the cerebrospinal fluid | baseline and 6 months
  Lipid levels

CONTACTS AND LOCATIONS:
Overall Officials: Florian Eichler, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be stored in a computer data repository at the Massachusetts General Hospital (MGH) Neurological Clinical Research Institute (NCRI). The purpose of this data repository is to capture and store data for clinical research. The repository will combine data from multiple studies. Datasets will be shared with researchers who want to advance understanding of Neurological Disease. These datasets will not contain any personal identifiable information.